CLINICAL TRIAL: NCT03655834
Title: Individualized Pemetrexed Dosing in Patients With Non-small Cell Lung Cancer or Mesothelioma Based on Renal Function to Improve Treatment Response
Brief Title: Dose Individualization of Pemetrexed - IMPROVE-III
Acronym: IMPROVE-III
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IMPROVE-III
Record Dates: First submitted 2018-05-14; First posted 2018-08-31 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Non Small Cell Lung Cancer; Mesothelioma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Mesothelioma | interventions — Pemetrexed; Clinical Trials, Phase I as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Microdosing (Experimental): Patients will be administered a microdose of pemetrexed with subsequent pharmacokinetic assessment. Afterwards the patients will continue in either IMPROVE-I or -II for second pharmacokinetic assessment
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed — patients will be administered a microdose with subsequent pharmacokinetic assessment.
  Other Names: Microdosing

SUMMARY:
Rationale:

Pemetrexed is a multi-targeted folate antagonist, which is primarily indicated for the treatment of advanced non-small cell lung cancer (NSCLC) and mesothelioma. Dosing of cytotoxic agents like pemetrexed requires balancing the dual risk of sub-therapy and toxicity. Administration of pemetrexed to patients with a creatinine clearance <45 ml/min is currently not advised. Pemetrexed is dosed based on body surface area (BSA), while renal function and dose are the sole determinants for systemic exposure. This causes 3 major issues:

1. In patients with renal dysfunction, BSA-based dosing may lead to haematological toxicity
2. Patients have to discontinue treatment due to declining renal function, and are withheld effective treatment
3. Even in patients with adequate renal function (GFR >45 ml/min) treatment may be improved by individualized dosing based on renal function, resulting in less toxicity. Also, BSA-based dosing may lead to ineffective therapy in patients with above average renal function.

The investigators aim to address these problems.

Objective: The overall main objective is to develop a safe and effective individualized dosing regimen for pemetrexed.

Study design: IMPROVE-III is an explorative microdosing study to assess the extrapolability of microdose-pharmacokinetics to the pharmacokinetics of a therapeutic dose.

Study population: IMPROVE-III includes 10 patients of IMPROVE-I and/or IMPROVE-II.

Intervention: patients will be administered a microdose with subsequent pharmacokinetic assessment.

Main study endpoints: The predictive performance of microdosing to predict full dose pharmacokinetics

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old
2. Planned for treatment with pemetrexed-based chemotherapy in IMPROVE-I or -II.
3. Eastern Cooperative Oncology Group (ECOG) performance score of 0-2
4. Subject is able and willing to sign the Informed Consent Form

Exclusion Criteria:

1. Conditions that affect haemostasis in a way that blood drawing is complicated (to be assessed by physician)
2. Contraindications for treatment with pemetrexed in line with the summary of product characteristics (SmPC) (except for creatinine clearance <45 ml/min in IMPROVE-I)

   1. Hypersensitivity to the active substance or to any of the excipients
   2. Pregnancy or lactation
   3. Concomitant yellow fever vaccine
3. The presence of clinically relevant pharmacokinetic interactions, according to the current SmPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
The predictive performance of microdosing to predict full dose pharmacokinetics | 3 months
  Mean relative prediction error (MPE)
The predictive performance of microdosing to predict full dose pharmacokinetics | 3 months
  Root mean squared relative prediction error (RMSE)
Exposure (AUC) after microdose | 1 day
  mg*h/l

CONTACTS AND LOCATIONS:
Overall Officials: Rob ter Heine, PhD, Principal Investigator — Radboud University Medical Center
Locations (5):
- Netherlands (5):
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - Antoni van Leeuwenhoek, Amsterdam
  - Maastricht University Medical centre, Maastricht
  - Radboud university medical centre, Nijmegen
  - Erasmus University Medical Centre, Rotterdam

REFERENCES:
- [Derived] Boosman RJ, de Rouw N, Huitema ADR, Burgers JA, Ter Heine R. Prediction of the pharmacokinetics of pemetrexed with a low test dose: A proof-of-concept study. Br J Clin Pharmacol. 2023 Feb;89(2):699-704. doi: 10.1111/bcp.15520. Epub 2022 Sep 21. PMID 36053283